CLINICAL TRIAL: NCT01042015
Title: Emergency Preservation and Resuscitation for Cardiac Arrest From Trauma
Brief Title: Emergency Preservation and Resuscitation (EPR) for Cardiac Arrest From Trauma
Acronym: EPR-CAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment was too slow with little potential for success. The complexities and resources needed for the intervention outweigh the very low probability of benefiting a rare patient. The DSMB and investigators agreed to terminate the study.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Samuel Tisherman, Professor of Surgery, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00062740
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrest From Trauma
Keywords: trauma; cardiac arrest; hemorrhagic shock
MeSH Terms: conditions — Wounds and Injuries; Heart Arrest; Shock, Hemorrhagic | interventions — Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Concurrent controls (Active Comparator): These subjects would undergo standard resuscitative efforts.
  Interventions: Other: Standard resuscitation
- Emergency preservation and resuscitation (Experimental): These subjects would undergo the complete EPR protocol, including rapid induction of hypothermia, resuscitative surgery, and resuscitation with cardiopulmonary bypass.
  Interventions: Combination Product: Emergency preservation and resuscitation

INTERVENTIONS:
Combination Product: Emergency preservation and resuscitation — This involves the induction of profound hypothermia using a flush of ice-cold saline into the aorta. Once hypothermia is achieved, the subject would undergo rapid operative interventions to control bleeding followed by resuscitation/rewarming with cardiopulmonary bypass.
  Arms: Emergency preservation and resuscitation
Other: Standard resuscitation — Standard resuscitation includes an emergency department thoracotomy, open cardiac massage, and fluid resuscitation.
  Arms: Concurrent controls

SUMMARY:
The goal of this study is to rapidly cool trauma victims who have suffered cardiac arrest from bleeding with a flush of ice-cold sodium chloride to preserve the patient to enable surgical control of bleeding, followed by delayed resuscitation with cardiopulmonary bypass.

DETAILED DESCRIPTION:
The intent of the technique to be studied is to induce a state of hypothermic preservation in trauma victims who have exsanguinated to the point of cardiac arrest. In appropriately selected subjects, after an initial emergency attempt at resuscitation with standard techniques, an arterial catheter will be inserted into the descending thoracic aorta. Using appropriate tubing, pump, and heat exchanger,a large quantity of ice-cold saline (0.9% Sodium Chloride for Injection USP) will be pumped as rapidly as possible into the aorta with the goal of cooling the brain (tympanic membrane temperature, Tty) to <10 C. If possible, a large venous catheter will be placed and recirculation of fluid established.

Once the subject has been sufficiently cooled, bleeding will be controlled surgically. The subject will then be resuscitated and rewarmed with full cardiopulmonary bypass.

The goal is to improve neurologically-intact survival in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Penetrating trauma with clinical suspicion of exsanguinating hemorrhage
* At least 1 sign of life at the scene (pulse, respiratory efforts, spontaneous movements, reactive pupils)
* Loss of pulse <5 min prior to Emergency Department (ED) arrival or in ED or operating room
* ED thoracotomy performed without immediate return of a palpable pulse in the carotid arteries after clamping the descending thoracic aorta

Exclusion Criteria:

* No signs of life for >5 min prior to the decision to initiate EPR
* Obvious non-survivable injury
* Suggestion of traumatic brain injury, such as significant facial or cranial distortion
* Electrical asystole
* Rapid external assessment of the injuries suggests massive tissue trauma or blunt trauma involving multiple body regions
* Pregnancy
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is survival to hospital discharge without major disability (Glasgow Outcome Scale-Extended >5). | Hospital discharge

SECONDARY OUTCOMES:
Feasibility of initiating EPR (cooling and achieving goal brain temperature) | 1 hour
Survival | 28 days
Neurologic functional outcome | 12 months
Multiple organ system dysfunction | During the initial hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Tisherman, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tisherman SA, Alam HB, Rhee PM, Scalea TM, Drabek T, Forsythe RM, Kochanek PM. Development of the emergency preservation and resuscitation for cardiac arrest from trauma clinical trial. J Trauma Acute Care Surg. 2017 Nov;83(5):803-809. doi: 10.1097/TA.0000000000001585. PMID 28538639

DOCUMENTS (1):
  • Study Protocol (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT01042015/Prot_000.pdf